CLINICAL TRIAL: NCT02975882
Title: A Phase 1 Study of ABI-009 (NAB-RAPAMYCIN) in Pediatric Patients With Recurrent or Refractory Solid Tumors, Including CNS Tumors as a Single Agent and in Combination With Temozolomide and Irinotecan
Brief Title: Nanoparticle Albumin-Bound Rapamycin, Temozolomide, and Irinotecan Hydrochloride in Treating Pediatric Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1514; NCI-2016-01412 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1514; ADVL1514 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1514 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2016-11-15; First posted 2016-11-29 (Estimated); Results first posted 2023-03-30 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Childhood Solid Neoplasm; Recurrent Malignant Solid Neoplasm; Recurrent Primary Central Nervous System Neoplasm; Refractory Malignant Solid Neoplasm; Refractory Primary Central Nervous System Neoplasm
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nab-rapamycin, temozolomide, irinotecan) (Experimental): Patients receive nanoparticle albumin-bound rapamycin IV over 30 minutes on days 1 and 8 beginning on cycle 1. Patients also receive temozolomide PO and irinotecan hydrochloride PO on days 1-5 beginning on cycle 2. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Sirolimus Albumin-bound Nanoparticles; Drug: Temozolomide

INTERVENTIONS:
Drug: Irinotecan Hydrochloride — Given PO
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; CPT11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U 101440E; U-101440E; U101440E
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Sirolimus Albumin-bound Nanoparticles — Given IV
  Other Names: ABI 009; ABI-009; ABI009; Albumin-bound Sirolimus; Fyarro; Nab-Rapamycin; Nab-sirolimus; Nanoparticle Albumin-Bound Rapamycin; Nanoparticle Albumin-bound Sirolimus; Sirolimus Albumin-bound Particles; Sirolimus Protein-bound Particles
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase I trial studies the side effects and best dose of nanoparticle albumin-bound rapamycin when given together with temozolomide and irinotecan hydrochloride in treating pediatric patients with solid tumors that have come back after treatment and a period of time during which the tumor could not be detected or has not responded to treatment. Nanoparticle albumin-bound rapamycin may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as temozolomide and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nanoparticle albumin-bound rapamycin, temozolomide, and irinotecan hydrochloride may cause the cancer to stop growing or shrink for a period of time and may lessen the symptoms that are caused by the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of nanoparticle albumin-bound rapamycin (ABI-009) administered as an intravenous infusion over 30 minutes on days 1 and 8 of a 21-day cycle, in combination with temozolomide and irinotecan hydrochloride (irinotecan) (administered on days 1-5) in pediatric patients with recurrent or refractory solid tumors, including central nervous system (CNS) tumors.

II. To define and describe the toxicities of single-agent ABI-009 administered as an intravenous infusion over 30 minutes on days 1 and 8 of a 21-day cycle in pediatric patients with recurrent or refractory solid tumors, including CNS tumors.

III. To define and describe the toxicities of ABI-009 administered as an intravenous infusion over 30 minutes on days 1 and 8 of a 21-day cycle in combination with temozolomide and irinotecan (administered on days 1-5) in pediatric patients with recurrent or refractory solid tumors, including CNS tumors.

IV. To characterize the pharmacokinetics of ABI-009 in pediatric patients with recurrent or refractory solid tumors, including CNS tumors.

SECONDARY OBJECTIVE:

I. To preliminarily define the antitumor activity of ABI-009 in combination with temozolomide and irinotecan within the confines of a phase 1 study.

EXPLORATORY OBJECTIVE:

I. To assess the biologic activity of ABI-009 by examining S6K1 and 4E-BP1 expression status in archival tumor tissue from solid tumor pediatric patients using immunohistochemistry.

OUTLINE: This is a dose-escalation study of nanoparticle albumin-bound rapamycin.

Patients receive nanoparticle albumin-bound rapamycin intravenously (IV) over 30 minutes on days 1 and 8 beginning on cycle 1. Patients also receive temozolomide orally (PO) and irinotecan hydrochloride PO on days 1-5 beginning on cycle 2. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a body surface area (BSA) of >= 0.2 m^2 at the time of study enrollment
* Patients with recurrent or refractory solid tumors, including CNS tumors, are eligible; patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG)
* Patients must have either measurable or evaluable disease
* Patient's current disease state must be one for which there is no known curative therapy
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age

  * Note: Neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the numerical eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately
* Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment

  * >= 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
* Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment
* Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
* Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair and the study-assigned research coordinator
* Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
* Stem cell infusions (with or without total body irradiation [TBI]):

  * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion (DLI) or boost infusion: >= 84 days after infusion, and no evidence of graft-versus-host disease (GVHD)
  * Autologous stem cell infusion including boost infusion: >= 42 days
* Cellular therapy: >= 42 days after the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
* X ray (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation
* Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131 iodine metaiodobenzylguanidine [131I-MIBG]): >= 42 days after systemically administered radiopharmaceutical therapy
* Irinotecan, temozolomide and mammalian target of rapamycin (mTOR) inhibitor exposure:

  * Patients who have received prior single agent therapy with irinotecan, temozolomide, or an mTOR inhibitor, excluding ABI-009, are eligible
  * Patients who have received prior therapy with ABI-009 are not eligible
  * Patients who have previously received irinotecan and temozolomide in combination without progressive disease while on therapy are eligible
  * Patients who have previously received irinotecan and temozolomide in combination and had significant toxicity with these two drugs are not eligible
  * Patients who have received prior therapy with all three agents in combination (i.e. irinotecan, temozolomide, and an mTOR inhibitor) are not eligible
* Adequate Bone Marrow Function Defined as:
* For patients with solid tumors without known bone marrow involvement (no older than 7 days at the start of therapy):

  * Peripheral absolute neutrophil count (ANC) >= 1000/mm^3
  * Platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
  * Hemoglobin >= 8.0 g/dl at baseline (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows (no older than 7 days at the start of therapy):

  * Age: maximum serum creatinine (mg/dL)
  * 1 to < 2 years: 0.6 (male and female)
  * 2 to < 6 years: 0.8 (male and female)
  * 6 to < 10 years: 1 (male and female)
  * 10 to < 13 years: 1.2 (male and female)
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age (no older than 7 days at the start of therapy)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x ULN = 135 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L (no older than 7 days at the start of therapy)
* Serum albumin >= 2 g/dL (no older than 7 days at the start of therapy)
* Pulse oximetry > 94% on room air if there is clinical indication for determination (e.g. dyspnea at rest)
* Patients with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants and well controlled
* Nervous system disorders (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0) resulting from prior therapy must be =< grade 2 with the exception of decreased tendon reflex (DTR); any grade of DTR is eligible
* Serum triglyceride level =< 300 mg/dL (no older than 7 days at the start of therapy)
* Serum total cholesterol level =< 300 mg/dL (no older than 7 days at the start of therapy)
* Random or fasting blood glucose =< the upper normal limits for age; if the initial blood glucose is a random sample that is outside of the normal limits, then follow-up fasting blood glucose can be obtained and must be =< the upper normal limits for age (no older than 7 days at the start of therapy)
* International normalized ratio (INR) =< 1.5 (no older than 7 days at the start of therapy)
* Not currently receiving anticoagulation therapy
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Tissue blocks or slides must be sent for all patients; if tissue blocks or slides are unavailable, the study chair must be notified prior to enrollment

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies; pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method both during and for 6 months after participation in this study; abstinence is an acceptable method of contraception
* Patients receiving corticosteroids must have been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients must not have received enzyme-inducing anticonvulsants for at least 7 days prior to enrollment
* Patients who are currently receiving therapeutic anticoagulants (including aspirin, low molecular weight heparin, and others) are not eligible
* Patients must not be receiving any strong CYP3A4 or P-glycoprotein (P-gp) inducers or inhibitors within 7 days prior to enrollment; moderate inducers or inhibitors of CYP3A4 and P-gp should also be avoided during ABI-009 treatment, if possible
* Patients with interstitial lung disease and/or pneumonitis are not eligible
* Patients with a history of allergic reactions attributed to compounds of similar composition, including macrolide and ketolide antibiotics, temsirolimus/other mTOR inhibitors, temozolomide or irinotecan are not eligible
* Patients with hypersensitivity to albumin are not eligible
* Patients who have had or are planning to have the following invasive procedures are not eligible:

  * Major surgical procedure, laparoscopic procedure, open biopsy or significant traumatic injury within 28 days prior to enrollment
  * Subcutaneous port placement or central line placement is not considered major surgery; external central lines must be placed at least 3 days prior to enrollment and subcutaneous ports must be placed at least 7 days prior to enrollment
  * Core biopsy within 7 days prior to enrollment
  * Fine needle aspirate within 7 days prior to enrollment
  * NOTE: For purposes of this study, bone marrow aspirate and biopsy are not considered surgical procedures and therefore are permitted within 14 days prior to start of protocol therapy
* Patients with current deep vein thrombosis or deep vein thrombosis within the past 6 months are not eligible
* Patients with a history of, or current grade 4 depression are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who have known bone marrow involvement are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart L Cramer, Principal Investigator — COG Phase I Consortium
Locations (21):
- United States (21):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Cramer SL, Reddy AT, Minard CG, Voss S, Fox E, Liu X, Denic K, Reid JM, Weigel BJ. A Phase 1 Study of ABI-009 (Nab-sirolimus) in Combination With Temozolomide and Irinotecan in Pediatric Patients With Recurrent or Refractory Solid Tumors, Including CNS Tumors-A Children's Oncology Group Pediatric Early Phase Clinical Trial Network Study ADVL1514. Cancer Med. 2024 Nov;13(21):e70376. doi: 10.1002/cam4.70376. PMID 39487711

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum Cohort With Dose Level 1: 35 mg/m^2 ABI-009 + 90 mg/m^2 Irinotecan + 125 mg/m^2 Temozolomide
- Stratum Cohort With Dose Level -1: 20 mg/m^2 ABI-009 + 90 mg/m^2 Irinotecan + 125 mg/m^2 Temozolomide
- Stratum Cohort With Dose Level -2; PK Cohort With Dose Level -2: 15 mg/m^2 ABI-009 + 90 mg/m^2 Irinotecan + 125 mg/m^2 Temozolomide
Period: Overall Study
Arm/Group | Stratum Cohort With Dose Level 1 | Stratum Cohort With Dose Level -1 | Stratum Cohort With Dose Level -2 | PK Cohort With Dose Level -2
Started | 5 | 13 | 9 | 6
Completed | 1 | 0 | 0 | 0
Not Completed | 4 | 13 | 9 | 6
Not completed — Adverse Event | 1 | 2 | 1 | 1
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 3 | 7 | 4 | 3
Not completed — Physician Decision | 0 | 2 | 4 | 2
Not completed — Ineligible | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients must have a body surface area (BSA) of >= 0.2 m^2 at the time of study enrollment: Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum Cohort With Dose Level 1 | Stratum Cohort With Dose Level -1 | Stratum Cohort With Dose Level -2 | PK Cohort With Dose Level -2 | Total
Number analyzed (Participants) | 5 | 13 | 9 | 6 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 10 | 8 | 6 | 28
  Between 18 and 65 years | 1 | 3 | 1 | 0 | 5
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 11 [7 to 20] | 13 [3 to 20] | 12 [1 to 21] | 8 [2 to 16] | 12 [1 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 2 | 10
  Male | 2 | 11 | 6 | 4 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 5 | 10 | 8 | 5 | 28
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 5
  White | 4 | 6 | 5 | 3 | 18
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 4 | 1 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Cycle 1 and 2 Dose Limiting Toxicities Attributable to Nanoparticle Albumin-bound Rapamycin
Description: Number of patients with cycle 1 and 2 dose limiting toxicities possibly, probably, or definitely attributable with nanoparticle albumin-bound rapamycin stratified by dose level.
Time Frame: Up to 42 days
Population: All DLT evaluable Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum Cohort With Dose Level 1 | Stratum Cohort With Dose Level -1 | Stratum Cohort With Dose Level -2 | PK Cohort With Dose Level -2
Number analyzed (Participants) | 5 | 6 | 6 | 4
Participants | 1 | 2 | 1 | 1

2. Primary Outcome: Number of Patients With Adverse Events
Description: The number of patients with adverse events that are at least possibly attributable to nanoparticle albumin-bound rapamycin stratified by dose level.
Time Frame: Up to 24 months
Population: All Eligible Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum Cohort With Dose Level 1 | Stratum Cohort With Dose Level -1 | Stratum Cohort With Dose Level -2 | PK Cohort With Dose Level -2
Number analyzed (Participants) | 5 | 12 | 9 | 6
Participants | 4 | 12 | 8 | 5

3. Primary Outcome: Area Under the Serum of Nanoparticle Albumin-bound Rapamycin Concentration Curve
Description: Median with minimum and maximum values of the area under the drug concentration over time curve stratified by dose level.
Time Frame: Days 1, 2, 3, 4, and 8
Population: All Eligible Patients
Measure: Mean (Full Range); unit: hr*ng/mL
Arm/Group | Stratum Cohort With Dose Level 1 | Stratum Cohort With Dose Level -1 | Stratum Cohort With Dose Level -2 | PK Cohort With Dose Level -2
Number analyzed (Participants) | 5 | 12 | 9 | 6
hr*ng/mL | 13654 [8610.0 to 19617.0] | 9532 [5352.0 to 18625.0] | 8666 [5074.0 to 12224.0] | 7988.5 [4826.0 to 11366.0]

4. Secondary Outcome: Number of Patients With Antitumor Activity of Nanoparticle Albumin-bound Rapamycin
Description: The number of response-evaluable patients with best overall response of complete response (CR), disappearance of all target lesions; or partial response (PR), >=50% decrease in the sum of the products of the two perpendicular diameters of all target lesions (up to 5), while on study therapy stratified by dose level; Overall response (OR)=CR+PR.
Time Frame: Up to 24 months
Population: All Eligible Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum Cohort With Dose Level 1 | Stratum Cohort With Dose Level -1 | Stratum Cohort With Dose Level -2 | PK Cohort With Dose Level -2
Number analyzed (Participants) | 5 | 12 | 9 | 6
Participants | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Stratum Cohort With Dose Level 1 | Stratum Cohort With Dose Level -1 | Stratum Cohort With Dose Level -2 | PK Cohort With Dose Level -2
All-Cause Mortality (participants affected / at risk) | 0/5 | 2/12 | 1/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 4/5 | 12/12 | 8/9 | 5/6
Other Adverse Events (participants affected / at risk) | 5/5 | 12/12 | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum Cohort With Dose Level 1 (N=5) | Stratum Cohort With Dose Level -1 (N=12) | Stratum Cohort With Dose Level -2 (N=9) | PK Cohort With Dose Level -2 (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 4 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Delayed puberty (Endocrine disorders) | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 3 | 0
Gastrointestinal disorders - Other, Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gum infection (Infections and infestations) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 2 | 1 | 1
Hypertension (Vascular disorders) | 2 | 2 | 4 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 3 | 6 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 1 | 4 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial tamponade (Cardiac disorders) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 2 | 3 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Surgical and medical procedures - Other, RENAL STENT PLACEMENT (Surgical and medical procedures) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1 | 0 | 0
Urine output decreased (Investigations) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Weight gain (Investigations) | 0 | 0 | 1 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
White blood cell decreased (Investigations) | 2 | 1 | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum Cohort With Dose Level 1 (N=5) | Stratum Cohort With Dose Level -1 (N=12) | Stratum Cohort With Dose Level -2 (N=9) | PK Cohort With Dose Level -2 (N=6)
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 4 | 3 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 6 | 6 | 3
Alkaline phosphatase increased (Investigations) | 2 | 3 | 3 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 2 | 1
Anal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 11 | 8 | 5
Anorexia (Metabolism and nutrition disorders) | 5 | 8 | 7 | 4
Anxiety (Psychiatric disorders) | 2 | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 5 | 5 | 3
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 3 | 2
Bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 1 | 0
Blurred vision (Eye disorders) | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 2 | 2 | 2 | 0
Cholesterol high (Investigations) | 3 | 3 | 8 | 4
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 8 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 2
Creatinine increased (Investigations) | 1 | 3 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 3 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 4 | 5 | 3
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1
Edema face (General disorders) | 2 | 0 | 0 | 0
Edema limbs (General disorders) | 1 | 1 | 1 | 0
Endocrine disorders - Other, (Endocrine disorders) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Eye disorders - Other, Double vision (Eye disorders) | 0 | 0 | 0 | 1
Eye disorders - Other, Left eye itching (Eye disorders) | 0 | 0 | 0 | 1
Eye disorders - Other, RIGHT ESOTROPIA (Eye disorders) | 1 | 0 | 0 | 0
Eye disorders - Other, visual disturbance (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 5 | 9 | 7 | 3
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fever (General disorders) | 1 | 4 | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Flashing lights (Eye disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 2 | 1 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, Lip Lesion (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, MOTILITY (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorders - Other, hematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, (General disorders) | 0 | 1 | 0 | 0
General disorders and administration site conditions - Other, LEFT SIDE HEMIPARESIS (General disorders) | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Genital edema (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 4 | 1
Hematuria (Renal and urinary disorders) | 2 | 3 | 3 | 2
Hemoglobin increased (Investigations) | 1 | 0 | 0 | 0
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hepatobiliary disorders - Other, (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3 | 8 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 4 | 1 | 2 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 4 | 2 | 6 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 | 4 | 5 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 6 | 5 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 5 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 3 | 5 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 6 | 7 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 5 | 5 | 1
Hypotension (Vascular disorders) | 2 | 1 | 2 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
INR increased (Investigations) | 0 | 1 | 1 | 0
Immune system disorders - Other, SEASONAL ALLERGIES (Immune system disorders) | 1 | 0 | 0 | 0
Infections and infestations - Other, (Infections and infestations) | 0 | 1 | 0 | 0
Infections and infestations - Other, C. DIFF (Infections and infestations) | 0 | 1 | 0 | 0
Infections and infestations - Other, COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3 | 3 | 0
Investigations - Other, (Investigations) | 0 | 1 | 0 | 0
Investigations - Other, AFP Tumor Marker Increase (Investigations) | 0 | 0 | 0 | 1
Investigations - Other, BICARBONATE < LLN (Investigations) | 1 | 0 | 0 | 0
Investigations - Other, C-reactive protein increased (Investigations) | 0 | 0 | 1 | 1
Investigations - Other, DECREASED CARBON DIOXIDE (Investigations) | 1 | 0 | 0 | 0
Investigations - Other, HDL Cholesterol decreased (Investigations) | 0 | 0 | 0 | 1
Investigations - Other, HYPOCHLOREMIA (Investigations) | 0 | 1 | 0 | 0
Investigations - Other, Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 1 | 1 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 0
Lipase increased (Investigations) | 3 | 1 | 1 | 0
Localized edema (General disorders) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 4 | 6 | 7 | 4
Malaise (General disorders) | 2 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 2 | 0 | 0
Metabolism and nutrition disorders - Other, HYPOCHLOREMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Metabolism and nutrition disorders - Other, Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle weakness right-sided (Nervous system disorders) | 0 | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, toe pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 10 | 6 | 4
Neck edema (General disorders) | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Nervous system disorders - Other, Disconjugated gaze (Nervous system disorders) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 3 | 3 | 7 | 2
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Oculomotor nerve disorder (Nervous system disorders) | 1 | 1 | 0 | 0
Oral dysesthesia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 3 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 4 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1
Periorbital edema (Eye disorders) | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Phantom pain (Nervous system disorders) | 0 | 2 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 5 | 9 | 7 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 4 | 4 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Renal and urinary disorders - Other, (Renal and urinary disorders) | 0 | 0 | 1 | 0
Reproductive system and breast disorders - Other, (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea and Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 1 | 0 | 0
Serum amylase increased (Investigations) | 1 | 1 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 5 | 7 | 4
Skin and subcutaneous tissue disorders - Other, ATOPIC DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Diaper rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Skin erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, bug bite (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, forehead abrasion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 2 | 1 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Spasticity (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 3 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 7 | 6 | 3
Weight gain (Investigations) | 1 | 1 | 2 | 0
Weight loss (Investigations) | 4 | 5 | 5 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
White blood cell decreased (Investigations) | 4 | 6 | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/82/NCT02975882/Prot_SAP_000.pdf